CLINICAL TRIAL: NCT01090375
Title: Regulation of Intraarticular and Synovium-related Biomarkers of Osteoarthritis. Effect of Acute Mechanical Joint Loading
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Danish Rheumatism Association (Other); Danish Ministry of Health, Internal Affairs (Unknown); Danish National Research Council (Unknown); The Danish Medical Research Council (Other)
Model: Parallel | Purpose: Basic Science
Other Study IDs: H-KF-306126
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Osteoarthritis; Exercise
Keywords: osteoarthritis; biochemical markers; cartilage; inflammation; microdialysis
MeSH Terms: conditions — Osteoarthritis; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Exercise
- Non Exercise (Placebo Comparator)
  Interventions: Other: Non Exercise

INTERVENTIONS:
Other: Exercise
  Arms: Exercise
Other: Non Exercise
  Arms: Non Exercise

SUMMARY:
In the present study the microdialysis method is used to investigate biochemical changes within and around the joint simultaneously in both the resting state and in a joint that had been subjected to exercise. The aim of the present study was, by applying the microdialysis technique, to monitor markers of cartilage breakdown and inflammation in 2 different positions of the knee (inside and in the inner part of the knee capsule) in a group of human females with knee osteoarthritis over a period of 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* verified osteoarthritis (x-ray)of the knee, female,

Exclusion Criteria:

* dementia, inflammatory diseases, regular pain medication

Ages: 55 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Dates: Start 2008-08; Primary Completion 2009-03 (Actual)

REFERENCES:
- [Derived] Helmark IC, Mikkelsen UR, Borglum J, Rothe A, Petersen MC, Andersen O, Langberg H, Kjaer M. Exercise increases interleukin-10 levels both intraarticularly and peri-synovially in patients with knee osteoarthritis: a randomized controlled trial. Arthritis Res Ther. 2010;12(4):R126. doi: 10.1186/ar3064. Epub 2010 Jul 1. PMID 20594330